CLINICAL TRIAL: NCT06817005
Title: Feasibility Study of the Nociception Level (NOL) Index for Intraoperative Assessment of Nociception During Cardiac Surgery
Brief Title: Nociception Monitoring During Cardiac Surgery
Acronym: MoNOLcard
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9529
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-01

CONDITIONS: Nociception; NOL Index; Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): nociception monitor device for intraoperative nociception monitoring during cardiac surgery.
  Interventions: Device: Intervention arm

INTERVENTIONS:
Device: Intervention arm — Prior to general anesthesia induction, a finger is inserted into the probe which is connected to the PMD200® to provide the NOL index. This output, a single dimensionless number from 0 to 100, correlated proportionally to nociception.

SUMMARY:
Cardiac surgery is frequently a source of acute or chronic pain. According to the International Association for the Study of Pain (IASP), nociception is defined as "the neural mechanisms of encoding and processing harmful stimuli," while pain is defined as "an undesirable sensory and emotional experience associated with real tissue damage". When patients are under general anesthesia (GA) during surgery, a lack of intraoperative analgesia can expose them to high levels of pain sensitization associated with surgical nociceptive stimuli. The response to the surgical nociceptive stress (via activation of the autonomic nervous system) can lead to alterations in hemodynamic or metabolic status, coagulation or the immune system. In addition, it is now well established that acute intra- and post-operative pain is directly related to the onset of chronic pain, particularly in the post-sternotomy period. On the contrary, excessive administration of opioid analgesics causes moderate to severe side effects (nausea, vomiting, bradypnea, delayed awakening, prolongation of recovery time, hyperalgesia syndrome, postoperative tolerance to opioids leading to misuse or occurrence of DCPO), which will result in postoperative morbidity for the patient independent of the surgery. Indeed, in cardiac surgery, there is a dose-dependent relationship between the intraoperative use of opioid analgesics such as remifentanil and the occurrence of postoperative hyperalgesia. The interest in intraoperative monitoring of nociception has therefore clearly increased in order to improve patient care from the point of view of intra- and postoperative pain management: administering a sufficient and personalized dose of analgesics, neither too high nor too low.

Strategies to prevent perioperative pain must therefore be developed to avoid sensitizing the patient to pain and thus limiting the onset of CD, or conversely, to avoid the onset of side effects from excessive analgesic treatment. These strategies include intra-operative pain monitoring. Numerous medical devices are available on the market to measure the level of nociception in patients undergoing GA. The vast majority of these monitors analyse clinical parameters that assess the balance between the sympathetic and parasympathetic nervous systems. Of all the monitors available, there is currently only one multiparametric monitor, the PMD200® which provides the Nociception Level Index or NOL Index (Medasense, Ramat Gan, Israel). In fact, the latter incorporates 5 parameters in its assessment of nociception: heart rate, RR segment variability, pulse wave amplitude, skin conductance level and skin temperature with the number of variations of these last two parameters. New devices for monitoring nociception used in the administration of intraoperative intravenous opioid agents could help to adjust the analgesia/nociception balance. In non-cardiac surgery, the NOL index has shown better sensitivity and specificity than variations in heart rate and blood pressure in detecting and helping to manage a surgical nociceptive stimulus during GA. This monitor has also enabled a dramatic reduction in the doses of intraoperative opioids administered.

In this study we hypothesized that monitoring of nociception using the NOL index is feasible during coronary artery surgery despite extracorporeal circulation.

ELIGIBILITY:
Inclusion criteria:

* adult patients
* patients undergoing on-pump cardiac surgery
* specific cardiac procedure : coronary artery bypass grafting

Exclusion criteria:

* patients with preoperative cardiac arrhythmia
* patients with a cardiac pacemaker
* emergency cardiac surgical procedure
* peripheral artery disease stage 2
* patients in shock prior to the cardiac surgery : mean arterial pressure 65mmHg with vasopressors
* persons participating in another interventional research
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The main evaluation criterion will be the NOL monitor signal loss time (loss of NOL digit display on the monitor screen) in relation to the total surgery time. Loss-of-signal and surgery times will be measured in minutes. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie Réanimation Cardiovasculaire, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No